CLINICAL TRIAL: NCT04224844
Title: Ultrasound-Guided Spinae Plane Block for Perioperative Pain Control in Carotid Endarterectomy.
Brief Title: Erector Spinae Plane Block for Carotid Endarterectomy
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: not recruiting, awaiting for changes in IRB
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AntalyaTRH029
Record Dates: First submitted 2020-01-07; First posted 2020-01-13 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spinae plane block group (Group 1) (Active Comparator): Patients will receive erector spinae plane block in addition to intravenous patient-controlled analgesia device containing tramadol.
  Interventions: Other: Erector spinae plane block
- Control group (Group 2) (Active Comparator): Control group will receive only intravenous patient-controlled analgesia device containing tramadol.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Erector spinae plane block — The block will be performed before the surgery. The spinous process of T2 or T3 wil be identified by an ultrasound guide, with the probe positioned longitudinally. A block needle will be inserted in the caudo-cephal direction. After the injection site is confirmed by 3 ml of physiological solution and correct position of the needle tip is confirmed, bupivacaine will be injected. The patients assigned to this group will also receive an intravenous patient-controlled analgesia device containing tramadol postoperatively.
  Arms: Erector spinae plane block group (Group 1)
Other: Control group — Control group will receive only patient-controlled analgesia device containing tramadol. No block will be performed.
  Arms: Control group (Group 2)

SUMMARY:
The purpose of this study is to test the hypothesis that erector spinae plane block will decrease intraoperative local anesthetic and postoperative analgesic consumption in patients undergoing carotid endarterectomy.

DETAILED DESCRIPTION:
Patients who decided to participate in the study will be randomized into 2 groups: Erector Spinae Plane Block Group (Group E) and Control Group (Group C). Intraoperative local anesthetic consumption, postoperative tramadol consumption, intraoperative and pain scores, hemodynamic parameters and patient satisfaction will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing carotid endarterectomy
* American Society of Anesthesiologists class 2 to 3
* Ability to consent

Exclusion Criteria:

* inability to communicate
* not understand the aim and objectives of the study
* not provide informed written consent
* contraindications for the block (local infection, coagulation disorders)
* hypersensitivity to the local anesthetics
* refusal of regional anesthesia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
24 hours tramadol consumption | 24 hours
  Total tramadol consumption in milligrams at 24 hrs will be scored.
6 hours tramadol consumption | 6 hours
  Total tramadol consumption in milligrams at 6 hrs will be scored.
12 hours tramadol consumption | 12 hours
  Total tramadol consumption in milligrams at 12 hrs will be scored.
Assesment of postoperative analgesia | 24 hours
  Post operative pain scores will be assessed using a numerical rating scala (NRS) (from 0=no pain, to10= worst pain imaginable) at 24 hrs.
Assesment of postoperative analgesia | 6 hours
  Post operative pain scores will be assessed using a numerical rating scala (NRS) (from 0=no pain, to10= worst pain imaginable) at 6 hours.
Assesment of postoperative analgesia | 12 hours
  Post operative pain scores will be assessed using a numerical rating scala (NRS) (from 0=no pain, to10= worst pain imaginable) at 12 hours.

SECONDARY OUTCOMES:
Amount of use of intraoperative local anesthetic. | 1 hour
  Intraoperative pain will be assessed using a visual analog scale (VAS) (from 0 = no pain to 10 = maximum possible pain). When intraoperative VAS is >3, supplemental local anesthetic will be administered to the surgical area by the surgeon. Amount of total local anesthetic in milligrams will be recorded at the end of the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Sait Kavakli, M.D., Principal Investigator — Antalya Training and Research Hospital
Locations (1):
- Antalya Training and Reseach Hospital, Antalya, Turkey (Türkiye)